CLINICAL TRIAL: NCT02920281
Title: Impact of Sleep Quality on Respiratory Function and Weaning of Mechanical Ventilation
Acronym: WEAN SLEEP 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: WEAN SLEEP 1
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Sleep Quality; Weaning of Mechanical Ventilation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

INTERVENTIONS:
Other: Polysomnography

SUMMARY:
The aim of the study is to evaluate the impact of sleep quality on the length of mechanical ventilation weaning, in intensive care unit patients

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation for at least 24 hours before the first weaning test
* difficult weaning of mechanical ventilation defined as failure to the first weaning test
* patients aged at least of 18 years

Exclusion Criteria:

* peripheral or central nervous system pathology
* known psychiatric pathology or agitation
* clinical worsening before polysomnography (shock with vasopressor drugs, coma with Glasgow scale < 8, PaO2/FiO2 ratio < 150 with respiratory distress signs)
* pregnant or breastfeeding women
* patient under legal guardianship or protection
* patient with no health insurance coverage
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Compare the length of weaning patients who have a poor quality of sleep to those who have a good quality sleep. | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, France

REFERENCES:
- [Derived] Thille AW, Reynaud F, Marie D, Barrau S, Rousseau L, Rault C, Diaz V, Meurice JC, Coudroy R, Frat JP, Robert R, Drouot X. Impact of sleep alterations on weaning duration in mechanically ventilated patients: a prospective study. Eur Respir J. 2018 Apr 19;51(4):1702465. doi: 10.1183/13993003.02465-2017. Print 2018 Apr. PMID 29519925